CLINICAL TRIAL: NCT06465225
Title: Prevention of Pressure Ulcers in Patients at Medium to High Risk of Pressure Ulcers Using the R'GO SOINS Overlay Mattress : Observational Study
Brief Title: Prevention of Pressure Ulcers in Patients at Medium to High Risk of Pressure Ulcers Using the R'GO SOINS Overlay Mattress
Acronym: PRESERVE
Status: Recruiting | Type: Observational
Sponsor: Nausicaa Medical (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A02335-40
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pressure Ulcer
Keywords: automated decompression air mattress; pressure ulcer; prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in nursing homes or long-stay geriatrics department
  Interventions: Device: Use of a powered alternating pressure air mattress

INTERVENTIONS:
Device: Use of a powered alternating pressure air mattress — Patients with a medium to high risk of developing pressure injury, without pressure injury, up during the day and lying between 15 and 20 hours per day will ly a on a R'GO Soins overlay mattress

SUMMARY:
The aim of the study is to determine the clinical value of using a powered alternating pressure air overlay mattress (P-APAM) in the prevention of pressure injury (PI) in patients at medium to high risk.

This study is noncomparative, observational study.

Patients older than 18 years of age, with a medium to high risk of PI, without PI, up during the day, and lying between 15 and 20 hours per day on a specific P-APAM will be included. The study will be conducted in nursing homes, and in long-stay geriatrics department.

Patients will be followed up for 35 days. The use of the P-APAM is associated with the usual PI prevention measures. The primary outcome is the percentage of patients who will develop at least one PI of at least stage 2 on the sacrum, spine, or heel between day 0 and day 35 . Secondary endpoints are patient assessments of comfort, caregiver satisfaction, mattress noise level, and mattress safety.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with a medium to high risk of developing pressure ulcers (clinical judgment and a score of [10 to 14] on the Braden scale (6 (maximum risk) to 23 (no risk))
* Patient without pressure injury on the day of inclusion
* Patient up during the day and lying down for more than 15 hours and less than 20 hours per day on an R'GO SOINS overlay mattress for less than 48 hours or since the day of inclusion
* Patient with a weight < 150kg
* Patient (or a trusted third party/legal representative) having been informed of the study and signing informed consent

Exclusion Criteria:

* Patient at end of life (estimated life expectancy less than 6 months)
* Patient discharge from the establishment expected within two months
* Patient already installed on an R'GO SOINS mattress topper for more than 48 hours before inclusion
* Patient with unstable spinal injury or other spinal disorder
* Patient with cervical or skeletal traction
* Patient with unstable spinal cord injury
* Patient with acute multiple trauma
* Patient with unstable posttraumatic bone fracture
* Participants will be excluded from the study if they meet the following combination of criteria indicative of malnutrition according to the 2021 French National Authority for Health guidelines (Participants must meet at least one phenotypic criterion and one etiological criterion to be considered malnourished and therefore ineligible for inclusion in the study) :

A) One or more of the following phenotypic criteria:

Significant unintentional weight loss: A weight loss of ≥ 5% within 1 month or ≥ 10% within 6 months Low Body Mass Index (BMI): BMI < 18.5 kg/m² for individuals under 70 years old, BMI < 21 kg/m² for individuals aged 70 years and older Reduced Muscle Mass Evident reduction in muscle mass AND

B) One of the following etiological criteria:

Inadequate nutritional intake:

Nutritional intake less than 50% of the energy requirements for more than one week Reduced food intake for more than two weeks Presence of Disease or Stress Metabolism Acute or chronic illness, or any condition causing metabolic stress that increases energy requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in nursing homes or long-stay geriatrics department
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who developed at least one stage 2 pressure injury | 35 days after installation on the mattress (at day 35)
  Percentage of patients who developed at least one stage 2 PI of the sacrum, backbone, or heel (areas of support when lying down)

SECONDARY OUTCOMES:
Percentage of patients who developed a o pressure injury (any stage), other than those of the sacrum, backbone, or heel between | 35 days after installation on the mattress (at day 35)
Assessment by the patient (or family or staff in the case of incapacity) of the comfort of the mattress (general comfort, stability) | 35 days after installation on the mattress (at day 35)
  On a scale from 0 (not satisfied at all) to 4 (very satisfied)
Assessment by the nursing staff with the use of the mattress (implementation, cleaning maintenance turning, changing to a sitting position) | 35 days after installation on the mattress (at day 35)
  On a scale from 0 (not satisfied at all) to 4 (very satisfied)
Assessment of the degree of maceration | 35 days after installation on the mattress (at day 35)
  On a scale from 1 (constantly moist) to 4 (rarely moist)
Assessment of mattress safety | At day 35
  By collecting any adverse event or mattress malfunction during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie MEAUME, PhD, Principal Investigator — Hôpital ROSCHILD
Locations (1):
- Multiples Facilities, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No